CLINICAL TRIAL: NCT06354036
Title: Transhiatal Tunnel Valvuloplasty for Reconstruction Following the Laparoscopic Proximal Gastrectomy，Phase II Trial
Brief Title: Transhiatal Tunnel Valvuloplasty for Reconstruction Following the Laparoscopic Proximal Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dong Bing Zhao, Clinical Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4465
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
Keywords: Proximal gastrectomy; Valvulopathy
MeSH Terms: conditions — Stomach Neoplasms; Heart Valve Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ThTV（the Transhiatal Tunnel Valvuloplasty technique group） (Experimental): Patients who meet the inclusion criteria will undergo ThTV anastomosis after proximal gastrectomy
  Interventions: Procedure: the Transhiatal Tunnel Valvuloplasty technique

INTERVENTIONS:
Procedure: the Transhiatal Tunnel Valvuloplasty technique — The ThTV esophagogastrostomy procedure involved placing a lengthy gastric tube into the lower mediastinum, firmly bound to the esophagus.

SUMMARY:
Patients who meet the inclusion criteria will undergo laparoscopic proximal gastric cancer radical surgery, and esophagogastric anastomosis will be performed using the ThTV method.

Review the surgical video and record the time for making the extracorporeal muscle flap, tunnel passage time, and anastomosis time. The production time of the muscle flap is based on the electric knife incision of the muscle flap as the starting point, and successfully penetrating the muscle flap as the endpoint. The tunnel passes through time, pulling the residual end of the esophagus, and starting to pass through the gastric muscle flap tunnel as the time starting point. The complete placement of the gastric tube into the lower mediastinum is used as the time endpoint. The anastomosis time is calculated from the first needle of suturing the residual stomach and the posterior wall of the esophagus until the end of the plasma flap suturing. Record perioperative indicators such as surgical time, bleeding volume, and postoperative hospital stay. The definition of anastomotic stenosis is that in gastroscopy, those who cannot pass through the anastomotic site with ultra-fine endoscopy are judged as anastomotic stenosis.

Postoperative pathology was performed using the 8th edition AJCC staging. Follow up every three months after surgery, including blood tests, liver and kidney function, and tumor markers. According to the situation, choose gastroscopy, upper gastrointestinal imaging, and chest abdominal pelvic enhanced CT. Evaluate postoperative reflux symptoms such as heartburn and sternal pain using the Visick grading system. Gastroscopy Los Angeles grading was used to evaluate postoperative reflux esophagitis.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed by gastroscopy pathological biopsy and imaging examination as early adenocarcinoma of the upper part of the stomach or adenocarcinoma of the esophageal gastric junction;
2. Tumor diameter<4cm, with no distant metastasis;
3. Clinical staging T1-3N0-1M0;
4. On the basis of proximal gastrectomy, 50% of the gastric volume can still be retained;
5. ECOG-PS status score 0-1 points (Eastern Cooperative Oncology Group).

Exclusion Criteria:

1. Patients undergoing preoperative neoadjuvant chemotherapy;
2. Patients with severe cardiovascular and pulmonary diseases who cannot tolerate laparoscopic surgery;
3. Incomplete clinical data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative reflux esophagitis | 1 year
  postoperative reflux

SECONDARY OUTCOMES:
the incidence of postoperative anastomotic fistula | 1 year
  Postoperative anastomotic fistula
the incidence of anastomotic stenosis | 1 year
  postoperative anastomotic stenosis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic and Gastric Surgical Oncology, National Cancer Center/ National Clinical Research for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No